CLINICAL TRIAL: NCT00564694
Title: Validation of an EORTC Quality of Life Questionnaire Module for Patients With Colorectal Cancer
Brief Title: Studying a Quality of Life Questionnaire in Patients With Colorectal Cancer
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Other Study IDs: CDR0000574769; EORTC-QLQ-CR29; EU-20783
Record Dates: First submitted 2007-11-27; First posted 2007-11-28 (Estimated); Last update posted 2013-10-29 (Estimated); Status verified 2009-08

CONDITIONS: Colorectal Cancer
Keywords: adenocarcinoma of the colon; recurrent colon cancer; stage I colon cancer; stage II colon cancer; stage III colon cancer; stage IV colon cancer; adenocarcinoma of the rectum; recurrent rectal cancer; stage I rectal cancer; stage II rectal cancer; stage III rectal cancer; stage IV rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Psychiatric Rehabilitation

INTERVENTIONS:
Procedure: psychosocial assessment and care
Procedure: quality-of-life assessment

SUMMARY:
RATIONALE: Collecting information about the quality of life of patients with colorectal cancer may help doctors learn more about the disease.

PURPOSE: This clinical trial is studying the European Organization of Research for the Treatment of Cancer (EORTC) quality-of-life-questionnaire in patients with colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* To test the reliability and clinical and psychometric validity of the European Organization of Research for the Treatment of Cancer (EORTC) quality of life questionnaire (QLQ-CR29) in an international sample of patients with colorectal cancer.

OUTLINE: This is a multicenter study. Patients are stratified into predetermined clinically distinct groups (colon cancer after surgery vs colon cancer undergoing adjuvant chemotherapy vs rectal cancer undergoing neoadjuvant radiotherapy vs rectal cancer after anterior resection with temporary stoma vs rectal cancer after abdominoperineal excision of rectum vs colorectal cancer undergoing palliative chemotherapy).

Quality-of-life data is collected alongside standard outcomes in patients undergoing treatment for colorectal cancer. Patients complete the European Organization of Research for the Treatment of Cancer (EORTC) quality of life questionnaire (QLQ-C30), the revised colorectal cancer module (QLQ-CR29), case report forms for clinical and sociodemographic data, and a debriefing questionnaire at different time points before, during, and after treatment. Some patients complete more sets of the same questionnaire at later time points to assess sensitivity to change over time and test-retest reliability. Reliability, and clinical and psychometric validity of the questionnaires are assessed by correlation analyses, exploration of known group comparisons, and responsiveness to clinical changes.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the colon or rectum
* No brain metastases or intracranial tumor extension with cognitive impairment

PATIENT CHARACTERISTICS:

* No limit on performance status
* Able to understand the language of the questionnaire
* No psychological, familial, sociological, or geographical condition potentially hampering compliance with the study protocol and follow-up schedule
* No other concurrent malignancies except basal cell carcinoma of the skin

PRIOR CONCURRENT THERAPY:

* No prior participation in this study (in a different subgroup)
* No concurrent participation in other quality of life studies that might interfere with this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2007-05; Primary Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Reliability and clinical and psychometric validity of the European Organization of Research for the Treatment of Cancer (EORTC) quality of life questionnaire (QLQ-CR29)

CONTACTS AND LOCATIONS:
Overall Officials: Jane Blazeby, MB, CHB, FRCS, BSc, MD, Study Chair — University Hospitals Bristol and Weston NHS Foundation Trust
Locations (5):
- Centre Alexis Vautrin, Vandœuvre-lès-Nancy, France
- Germany (2):
  - Charite University Medical Center of Berlin, Berlin
  - Klinikum der Universitaet Regensburg, Regensburg
- United Kingdom (2):
  - Basingstoke and North Hampshire NHS Foundation Trust, Basingstoke, England
  - Bristol Haematology and Oncology Centre, Bristol, England

REFERENCES:
- [Result] Arraras JI, Suarez J, Arias de la Vega F, Vera R, Asin G, Arrazubi V, Rico M, Teijeira L, Azparren J. The EORTC Quality of Life questionnaire for patients with colorectal cancer: EORTC QLQ-CR29 validation study for Spanish patients. Clin Transl Oncol. 2011 Jan;13(1):50-6. doi: 10.1007/s12094-011-0616-y. PMID 21239355
- [Result] Nowak W, Tobiasz-Adamczyk B, Brzyski P, Salowka J, Kulis D, Richter P. Adaptation of quality of life module EORTC QLQ-CR29 for Polish patients with rectal cancer: initial assessment of validity and reliability. Pol Przegl Chir. 2011 Sep;83(9):502-10. doi: 10.2478/v10035-011-0078-5. PMID 22166739
- [Result] Whistance RN, Conroy T, Chie W, Costantini A, Sezer O, Koller M, Johnson CD, Pilkington SA, Arraras J, Ben-Josef E, Pullyblank AM, Fayers P, Blazeby JM; European Organisation for the Research and Treatment of Cancer Quality of Life Group. Clinical and psychometric validation of the EORTC QLQ-CR29 questionnaire module to assess health-related quality of life in patients with colorectal cancer. Eur J Cancer. 2009 Nov;45(17):3017-26. doi: 10.1016/j.ejca.2009.08.014. Epub 2009 Sep 16. PMID 19765978